CLINICAL TRIAL: NCT07220304
Title: CaRi-Heart® Assessment of Risk and Evaluation of Inflammation in Coronary CT Angiography (CARE-CCTA): A Prospective U.S. Community-Based Study on the Impact of CaRi-Heart® Analysis in Patients Undergoing CCTA for Coronary Artery Disease
Brief Title: CaRi-Heart Assessment of Risk and Evaluation of Inflammation in Coronary CT Angiography (CARE-CCTA)
Acronym: CARE-CCTA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corazon Medical PC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CARE-CCTA-001
Record Dates: First submitted 2025-10-22; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Cardiovascular Inflammation
Keywords: CaRi-Heart; Coronary CT Angiography (CCTA); AI Cardiac Imaging; Coronary Inflammation; Cardiovascular Risk Stratification; Plaque Characterization; Community-Based Imaging; Noninvasive Cardiac Diagnostics; Artificial Intelligence in Cardiology
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Single-arm prospective diagnostic study evaluating the incremental value of CaRi-Heart® analysis in patients undergoing Coronary CT Angiography (CCTA) for suspected or known coronary artery disease
Masking Description: Open-label study. Both investigators and participants are aware of CaRi-Heart® analysis results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CaRi-Heart® Analysis Group (Experimental): Participants receiving standard CCTA with CaRi-Heart® software analysis to assess coronary inflammation and evaluate impact on clinical decision-making.
  Interventions: Device: CaRi-Heart® Analysis

INTERVENTIONS:
Device: CaRi-Heart® Analysis — CaRi-Heart® is an artificial-intelligence-based software device that analyzes coronary CT angiography (CCTA) images to quantify coronary inflammation and generate a CaRi-Heart Risk Score. The analysis provides color-coded visualization and quantitative metrics derived from perivascular fat tissue characteristics, enabling improved assessment of coronary artery disease risk.
  In this study, CaRi-Heart® analysis is applied prospectively to CCTA images obtained as part of standard clinical care. The results are reviewed by the interpreting physician and recorded to determine whether the additional information affects diagnostic interpretation or management decisions. No additional imaging, radiation, or contrast exposure occurs.
  Other Names: AI-based coronary inflammation analysis; CaRi-Heart Risk Score

SUMMARY:
This study evaluates the use of CaRi-Heart® analysis, an artificial-intelligence (AI) software tool that measures inflammation in the coronary arteries using images already captured during a standard Coronary CT Angiography (CCTA) exam. The goal is to determine whether the additional information provided by CaRi-Heart® changes clinical decision-making and helps improve early identification and management of coronary artery disease in community imaging centers. Patients who undergo CCTA as part of their regular care will be invited to have their scans analyzed using CaRi-Heart® at no extra cost, time, or radiation.

DETAILED DESCRIPTION:
This is a prospective, community-based interventional study designed to assess the incremental value of CaRi-Heart® analysis in patients undergoing Coronary CT Angiography (CCTA) for evaluation of suspected or known coronary artery disease.

CaRi-Heart® is a software-as-a-medical-device (SaMD) that uses advanced AI algorithms to quantify coronary inflammation and generate a CaRi-Heart® Risk Score from existing CCTA images. The analysis provides color-coded visualization and quantitative metrics that may improve risk stratification beyond traditional plaque and stenosis assessment.

The study aims to compare management decisions made before and after review of the CaRi-Heart® analysis, measuring how often the additional information influences diagnostic interpretation or changes treatment recommendations (such as preventive therapy or referral).

Approximately 15,000 participants will be enrolled across multiple outpatient imaging centers in Michigan. All data will be collected under standard clinical workflows with IRB approval, informed consent, and HIPAA compliance. No additional scanning, contrast, or radiation exposure will occur.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically indicated CCTA undertaken for evaluation of coronary artery disease.
2. Ability to provide written informed consent
3. Patient between 18 and 80 years old

Exclusion Criteria:

- 1. History of surgical revascularization (coronary artery bypass graft, CABG) 2. CCTA undertaken for structural heart disease evaluation (e.g. transcatheter aortic valve replacement (TAVR) 3. The CCTA is of poor quality or partly unanalysable due to artifacts, such as motion-artifacts, breathing-artifacts, stack-artifacts or blooming-artifacts.

4. Inability to provide required health information 5. Pregnancy or any known contraindication for CCTA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in clinical management decisions following CaRi-Heart® analysis | Up to 60 days following CCTA completion
  The proportion of patients for whom the addition of CaRi-Heart® analysis to standard Coronary CT Angiography (CCTA) results in a change in clinical management decisions, such as initiation or adjustment of preventive therapies (e.g., statins, antiplatelet agents, lifestyle modification, or cardiology referral).
  Management decisions before and after reviewing CaRi-Heart® results will be compared to quantify impact on diagnostic interpretation and treatment planning

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Corazon Imaging, Bay City, Michigan
  - Corazon Imaging, Berkley, Michigan
  - Corazon Imaging, Caro, Michigan
  - Corazon Imaging, Dearborn, Michigan
  - Corazon Imaging, Flint, Michigan
  - Corazon Imaging, Grand Rapids, Michigan
  - Corazon Imaging, Livonia, Michigan
  - Corazon Imaging, Macomb, Michigan
  - Corazon Imaging, Madison Heights, Michigan
  - Corazon Imaging, Mount Pleasant, Michigan
  - Corazon Imaging, Novi, Michigan
  - Corazon Imaging, Saginaw, Michigan
  - Corazon Imaging, Saint Clair Shores, Michigan
  - Corazon Imaging, Sterling Heights, Michigan
  - Corazon Imaging, Trenton, Michigan
  - Corazon Imaging, Waterford, Michigan
  - Corazon Imaging, Elizabethtown, Pennsylvania
  - Corazon Imaging, Lemoyne, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD) may be shared with qualified researchers upon reasonable request after study completion, subject to IRB approval, institutional policies, and a data-use agreement. Data elements may include demographic variables, CaRi-Heart® risk scores, and CCTA-derived imaging metrics. No protected health information (PHI) will be shared.